CLINICAL TRIAL: NCT04480411
Title: Use of Technology and Telemedicine to Improve Quality of Care in COVID 19 Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unavailable IT resources
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 56472
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Diagnoses Disease; Covid19
Keywords: Telemedicine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COVID-19 Patients (Experimental): Patients that are admitted to the hospital with COVID 19.
  Interventions: Behavioral: Doctorgram Patient Kit

INTERVENTIONS:
Behavioral: Doctorgram Patient Kit — Participants will use the Doctorgram Patient Kit for remote monitoring and remote use stethoscope.

SUMMARY:
The purpose of this study is to assess the use of technology including remote vital sign monitoring in improving quality of patient care, decreasing hospital admissions and re-admissions, decreasing hospital length of stay and decreasing use of personal protective equipment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient with COVID 19 or outpatient under investigation for or diagnosed with COVID 19
* Clinically stable (on 4L O2 or less, non ICU)
* Demonstrates ability to be trained in use of digital stethoscope technology

Exclusion Criteria:

* Pregnancy
* Delirium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Patient provider experience survey score | Once after completion of device use (up to 15 minutes to complete the survey)
  Five questions related to satisfaction with experience using home pulse oximetry, each on a scale of 1 (poor) to 5 (excellent) summed and averaged for an overall range of 1 to 5 (higher scores = better experience).
Provider experience survey score | Once after completion of device use (up to 15 minutes to complete the survey)
  Four questions related to satisfaction with experience using home pulse oximetry, each on a scale of 1 (poor) to 5 (excellent) summed and averaged for an overall range of 1 to 4 (higher scores = better experience).
Use of personal protective improvement | 6 months
  Level of personal protective improvement in an in-patient setting.
Number of in-patient encounters with COVID patients as a measure of provider exposure to high risk illness | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Parikh, MD, Principal Investigator — Stanford University; Julieta M Gabiola, MD, Principal Investigator — Stanford University; Nicholas Scoulios, MD, Principal Investigator — Stanford University; Lisa Shieh, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No